CLINICAL TRIAL: NCT02719340
Title: Short-segment Decompression and Reconstruction for Thoracolumbar Osteoporotic Fractures With Neurological Deficits: Clinical and Radiological Results of Minimum 2-year Follow-up
Brief Title: Short Segment Fixation in Thoracolumbar Osteoporotic Fracture
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Li Lin, Attending Physician, National Cheng-Kung University Hospital
Other Study IDs: SSF-TLF-103
Record Dates: First submitted 2016-02-18; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Spinal Fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: short segment fixation — posterior short-segment decompression and reconstruction (instrumentation on 1 level above and 1 level below the fractured vertebrae with posterolateral fusion)

SUMMARY:
Although long-segment posterior spinal fixation might provide more rigid fixation, the procedure increases perioperative morbidities in the elderly. The present study reviews the results of short-segment decompression and reconstruction in thoracolumbar fragile fractures.

DETAILED DESCRIPTION:
This study included 20 elderly patients with osteoporotic thoracolumbar burst fractures and neurological compromise. The participants were followed-up for a period of 40.6 (24-68) months. A visual analog scale (VAS) and the Oswestry Disability Index (ODI) were used to measure back pain and disability. Radiologic assessment and neurological status were also analyzed.

ELIGIBILITY:
Inclusion Criteria

* osteoporotic burst fracture at a single level of the thoracolumbar region
* dual-energy X-ray absorptiometry and T-score value less than -2.5

Exclusion Criteria

* translational displacement at the fracture site (fracture-dislocation)
* loss of structural integrity within the posterior osteoligamentous complex (such as flexion-distraction ligament disruption)
* spondylolisthesis of the adjacent vertebrae
* malignancy
* chronic steroid administration
* previous spinal surgery
* prior vertebroplasty and infection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty elderly patients (60-89 years, mean 73.2 years) with osteoporotic thoracolumbar burst fractures and neurological compromise
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | at least 2 years
  Functional outcome after surgery was evaluated using the Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Frankel's grade system | at least 2 years
  Frankel's grade system was used for assessment of neurologic function
Local kyphosis and vertebral wedge angle were measured as radiologic assessment (units of measure: degree) | at least 2 years
  Digital radiographs of the vertebral bodies were reviewed using the picture archiving and communication system (PACS).
anterior vertebral height | at least 2 years
  Measurements of the anterior vertebral height (AVH) ratio (% of normal)

IPD SHARING:
Plan to Share IPD: No